CLINICAL TRIAL: NCT05862688
Title: A Cohort Study on Anti-microbial Stewardship in PICU
Status: Not yet recruiting | Type: Observational
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: fdpicu-29
Record Dates: First submitted 2023-02-26; First posted 2023-05-17 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Infections
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Infection: patients with infection
  Interventions: Other: antimicrobial therapy
- non-infection: patients without infection

INTERVENTIONS:
Other: antimicrobial therapy — antimicrobial therapy
  Groups: Infection

SUMMARY:
Appropriate antimicrobial therapy is essential to ensuring positive patient outcomes. Inappropriate or suboptimal utilization of antibiotics can lead to increased length of stay, multidrug-resistant infections, and mortality. Critically ill intensive care patients are at risk of antibiotic failure and secondary infections associated with incorrect antibiotic use. Initiating effective therapy for infections based upon patients' risk factors, collection of appropriate cultures, daily evaluation of clinical status, and laboratory data, including antibiotic time outs, and shortened duration of therapy are ways to improve patients outcomes. Antimicrobial stewardship teams can assist ICU providers in managing and implementing these tactics. ICUs would benefit from employing empiric guidelines for antibiotic use, collecting appropriate specimens and implementing molecular diagnostics, optimizing the dosing of antibiotics, and reducing the duration of total therapy.

DETAILED DESCRIPTION:
Appropriate antimicrobial therapy is essential to ensuring positive patient outcomes. Inappropriate or suboptimal utilization of antibiotics can lead to increased length of stay, multidrug-resistant infections, and mortality. Critically ill intensive care patients are at risk of antibiotic failure and secondary infections associated with incorrect antibiotic use. Initiating effective therapy for infections based upon patients' risk factors, collection of appropriate cultures, daily evaluation of clinical status, and laboratory data, including antibiotic time outs, and shortened duration of therapy are ways to improve patients outcomes. Antimicrobial stewardship teams can assist ICU providers in managing and implementing these tactics. ICUs would benefit from employing empiric guidelines for antibiotic use, collecting appropriate specimens and implementing molecular diagnostics, optimizing the dosing of antibiotics, and reducing the duration of total therapy. This study conducted an antibiotic management cohort study in PICUs to discover the distribution of nosocomial infections in PICUs and to find controllable factors for the occurrence of nosocomial infections.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the ICU for more than 48 hour

Exclusion Criteria:

* Patients admitted to ICU less than 48 hours

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: ICU patient
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
survival rate | 21 days after ICU admission
  the survival rate of children in 21 days after ICU admission

SECONDARY OUTCOMES:
the length of ICU stay time | 21 days after ICU admission
  the length of ICU stay time

IPD SHARING:
Plan to Share IPD: No